CLINICAL TRIAL: NCT06268041
Title: Moderate-Intensity Exercise Versus High-Intensity Interval Training to Recover Walking Post-Stroke: HIT-Stroke Trial 2
Brief Title: HIT-Stroke Trial 2
Acronym: HST2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Kansas Medical Center (Other); University of Delaware (Other)
Responsible Party: Principal Investigator, Pierce Boyne, Associate Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 427659; R01HD093694 (NIH)
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Stroke
Keywords: gait; aerobic; locomotion
MeSH Terms: conditions — Stroke | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate-Intensity Aerobic Training (Active Comparator)
  Interventions: Behavioral: Moderate-Intensity Aerobic Training
- High-Intensity Interval Training (Experimental)
  Interventions: Behavioral: High-Intensity Interval Training

INTERVENTIONS:
Behavioral: Moderate-Intensity Aerobic Training — Overground and treadmill walking with speed continuously adjusted to maintain a target heart rate of 40 +/- 5% heart rate reserve, progressing up to 55 +/- 5% heart rate reserve.
  Arms: Moderate-Intensity Aerobic Training
Behavioral: High-Intensity Interval Training — Overground and treadmill walking with 30 second bursts at maximum speed alternated with 30-60 second passive recovery periods. Intended to achieve a target average heart rate above 60% heart rate reserve.
  Arms: High-Intensity Interval Training

SUMMARY:
People who had a stroke at least 6 months prior and who still have difficulty with walking will each be randomly assigned to receive either moderate or vigorous intensity walking exercise. Both protocols will be performed individually with a physical therapist for 45 minutes, 3x/week for 12 weeks. Measures including walking function will be assessed at baseline (PRE), after 4, 8 and 12 weeks of training (12WK) and at 3-month follow up (3moPOST), by raters who are unaware of the participant randomization.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-85 years at time of consenting
* Hemiparesis from ischemic and/or hemorrhagic strokes
* Most recent stroke for which participant sought treatment, at least 6 months prior to study consent
* Walking speed <1.0 m/s on the 10-meter walk test
* Able to walk 10m over ground with assistive devices as needed and no continuous physical assistance from another person (guarding and intermittent assistance for loss of balance allowed)
* Able to walk at least 3 minutes on the treadmill at ≥0.13m/s (0.3 mph)
* Stable cardiovascular condition (AHA class B, allowing for aerobic capacity <6 metabolic equivalents)
* Able to communicate with investigators, follow a 2-step command and correctly answer consent comprehension questions

Exclusion Criteria:

* Exercise testing uninterpretable for ischemia or arrhythmia (e.g. resting ECG abnormality that makes exercise ECG uninterpretable for ischemia and no other clinical testing from the past year available to rule out these conditions)
* Evidence of significant arrhythmia or myocardial ischemia on treadmill ECG graded exercise test in the absence of recent (past year) more definitive clinical testing (e.g. stress nuclear imaging) with negative result
* Hospitalization for cardiac or pulmonary disease within past 3 months
* Implanted pacemaker or defibrillator with an upper heart rate limit that would interfere with exercise testing or prescription, or with unknown limit
* Significant ataxia or neglect (score of 2 on NIH stroke scale item 7 or 11)
* Severe lower limb spasticity (Ashworth >2)
* Known recent history (<3 months) of unstable substance abuse or unstable mental illness
* Major post-stroke depression (Patient Health Questionnaire [PHQ-9] ≥ 10) in the absence of depression management by a health care provider
* Currently participating in physical therapy or another interventional study targeting walking function
* Recent (<2 weeks) or planned changes in lower limb orthotic or spasticity management
* Foot drop or lower limb joint instability without adequate stabilizing device, as assessed by a physical therapist
* Clinically significant neurologic disorder other than stroke or unable to walk outside the home prior to stroke
* Unable to walk outside the home prior to stroke
* Other significant medical condition likely to limit improvement or jeopardize safety as assessed by a physical therapist (e.g. joint contracture, gait limited by pain)
* Pregnancy
* Previous exposure to fast treadmill walking (>3 cumulative hours) in the past year

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2024-02-09 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
6-Minute Walk Test Distance | Change from Baseline to 12 weeks
  Total distance walked in 6 minutes in meters

SECONDARY OUTCOMES:
6-Minute Walk Test Distance | Change from Baseline to 3 month follow up
  Total distance walked in 6 minutes in meters
Self-Selected Gait Speed | Change from Baseline to 12 weeks
  From 10-meter walk test at self-selected speed, in meters per second
Fastest Gait Speed | Change from Baseline to 12 weeks
  From 10-meter walk test at fastest speed, in meters per second
PROMIS-Fatigue Scale version 8a | Change from Baseline to 3 month follow up
  An 8-item self-report questionnaire about symptoms of fatigue. Each item is rated from 1-5. Items are combined to obtain a total T score, where higher scores indicate greater fatigue.
Aerobic Capacity | Change from Baseline to 12 weeks
  Oxygen consumption rate at ventilatory threshold during treadmill graded exercise test, in milliliters per kilogram body mass per minute
EuroQol-5D-5L | Change from Baseline to 3 month follow up
  A 6-item questionnaire about quality of life, including: mobility, self-care, usual activities, pain/discomfort, anxiety/depression and overall health. Each item is scored from 1 to 5, where lower scores indicate greater quality of life. A total 'misery score' will be calculated by averaging the scores for each item.

CONTACTS AND LOCATIONS:
Overall Officials: Pierce Boyne, PT, DPT, PhD, Principal Investigator — University of Cincinnati
Locations (3):
- United States (3):
  - University of Delaware, Newark, Delaware
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Cincinnati, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Yes
The final, de-identified dataset and data documentation will be deposited into the Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Data and Specimen Hub (DASH) archive
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Will be submitted within one year of trial completion and will remain available indefinitely
Access Criteria: Established by the repository
URL: https://dash.nichd.nih.gov

REFERENCES:
- [Derived] Garrity C, Reisman DS, Billinger SA, Pressler D, Wagner E, Awosika O, Bartsch BL, Briton-Carpenter A, Carl D, Engler A, Foster J, Kim J, McCartney K, Moores A, Sucharew H, Thompson E, Walters K, Wasik E, Wright H, Yeazell M, Boyne P. Protocol for the HIT-Stroke Trial 2 randomized controlled trial: Moderate-intensity exercise versus high-intensity interval training to determine the optimal training intensity for walking rehabilitation in chronic stroke. medRxiv [Preprint]. 2025 Jul 31:2025.07.30.25332470. doi: 10.1101/2025.07.30.25332470. PMID 40766122

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-08-11): https://cdn.clinicaltrials.gov/large-docs/41/NCT06268041/SAP_000.pdf